CLINICAL TRIAL: NCT06578585
Title: Interventional, Randomized, Double-blind, Placebo-controlled Trial Investigating the Safety and Tolerability of Lu AG09222 When Coadministered With Ubrogepant in Participants With Migraine
Brief Title: A Trial Investigating Lu AG09222 With Ubrogepant in Participants With Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20527A
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ubrogepant with Lu AG09222 (Experimental): Participants will receive 2 doses of ubrogepant, then participants will receive Lu AG09222 followed by additional doses of ubrogepant.
  Interventions: Drug: Ubrogepant; Drug: Lu AG09222
- Ubrogepant with Placebo (Placebo Comparator): Participants will receive 2 doses of ubrogepant, then participants will receive placebo followed by additional doses of ubrogepant.
  Interventions: Drug: Ubrogepant; Drug: Placebo

INTERVENTIONS:
Drug: Ubrogepant — Tablet
Drug: Lu AG09222 — Solution for injection/infusion
  Arms: Ubrogepant with Lu AG09222
Drug: Placebo — Solution for injection/infusion
  Arms: Ubrogepant with Placebo

SUMMARY:
The main goal of this trial is to learn more about the safety and tolerability of Lu AG09222 when taken together with ubrogepant. This includes looking for any new or worsening medical issues the participants have with the treatment. During the trial, participants with migraine will receive ubrogepant oral tablets and an injection of either Lu AG09222 or a placebo.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine as defined by ICHD-3 guidelines confirmed at the Screening Visit.
* The participant has a history of migraine onset ≥12 months prior to the Screening Visit.
* The participant has ≥2 migraine days and headache occurring on <15 days per month for each month within the past 3 months prior to the Screening Visit.
* The participant has a body mass index (BMI) ≥18.5 and ≤ 35 kilograms per meter squared (kg/m^2) at the Screening Visit.

Exclusion Criteria:

* The participant has previously been dosed with an anti-pituitary adenylate cyclase-activating peptide (PACAP) treatment.
* The participant has participated in a clinical trial <30 days prior to the Screening Visit.
* The participant has taken any investigational medicinal product (IMP) <3 months or <5 half-lives of that product, whichever is longer, prior to Visit 1.
* The participant is pregnant, breastfeeding, intends to become pregnant, or is of childbearing potential and not willing to use adequate contraceptive methods.
* The participant has known or suspected hypersensitivity or intolerance to the IMP, auxiliary medicinal product (AxMP), or their excipients.

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to 92 Days

SECONDARY OUTCOMES:
AUC0-infinity: Area under the plasma concentration curve of ubrogepant from zero to infinity | Predose on Day 1 to Day 12
Cmax: maximum observed plasma concentration of ubrogepant | Predose on Day 1 to Day 12
tmax: nominal time corresponding to the occurrence of Cmax | Predose on Day 1 to Day 12
t½: apparent elimination half-life of ubrogepant | Predose on Day 1 to Day 12
Oral Clearance (CL/F) of ubrogepant | Predose on Day 1 to Day 12
Apparent volume of distribution (VZ/F) of ubrogepant | Predose on Day 1 to Day 12
Number of participants with anti-drug antibodies for Lu AG09222 | Up to 92 Days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (4):
- United States (4):
  - Clinical Neuroscience Solutions, Orlando, Florida
  - NeuroTrials Research, Atlanta, Georgia
  - Future Search Trials, Austin, Texas
  - Elevate Clinical Research, Seabrook, Texas